CLINICAL TRIAL: NCT02353676
Title: Bupivacaine For Postoperative Pain Control
Brief Title: Bupivacaine Supplementation For Postoperative Pain Control In Surgical Removal Of Mandibular Third Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cosmozone Dental Clinic (Other)
Responsible Party: Principal Investigator, pavan MANOHAR PATIL, DIRECTOR, Cosmozone Dental Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: COSMOZONE
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Anesthesia, Local
MeSH Terms: interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- BUPIVACAINE GROUP (Experimental): 1.5 ml of 0.5% Bupivacaine solution to be injected into the operative site postoperatively.
  Interventions: Drug: Bupivacaine
- PLACEBO GROUP (Placebo Comparator): 1.5 ml of saline solution to be injected into the opposite site postoperatively.
  Interventions: Other: SALINE

INTERVENTIONS:
Drug: Bupivacaine — 1.5 ml of 0.55 bupivacaine solution to be used as postoperative anesthetic agent for prolonged analgesia
  Other Names: ANAWIN
  Arms: BUPIVACAINE GROUP
Other: SALINE — 1.5 ml of placebo (saline solution) to be injected into the opposite site postoperatively.
  Arms: PLACEBO GROUP

SUMMARY:
Control of postoperative pain is a foremost goal in achieving a satisfactory postoperative recovery. Surgical removal of lower third molars is accompanied by postoperative pain that is at its peak in the first 12 hours. Our study evaluates if the use of 2% lidocaine hydrochloride for the surgical removal of lower third molars with a postoperative 0.5% bupivacaine supplementation would result in lesser postoperative pain and a decrease in ingestion of oral analgesics to control the pain when compared to a placebo.

DETAILED DESCRIPTION:
The study intends to enroll 100 patients [ASA 1] with bilateral symmetrical impacted mandibular third molars requiring surgical removal under local anesthesia. 2% Lidocaine hydrochloride with epinephrine bitartrate 1: 80000 in 3ml quantity will be utilized to achieve local anesthesia at the surgical site on both quadrants. Additional supplementation postoperative at the surgical site will be provided with either 1.5 ml of 0.5% bupivacaine with 1:80000 epinephrine solution or saline based on a split mouth randomized study design using a color and number coded envelop. All procedures will be performed by a single surgeon using a similar technique, under identical conditions at one month apart intervals. Pain scores will be assessed by the patient based on a 10cm Visual Analog Scale at intervals of 2, 4, 6, 12, 24, 36, 48, 72, 96 and 120 hours. The duration of soft tissue anesthesia postoperatively will be recorded by the patient. The number of analgesics ingested over 120 hours will be recorded by the patient. Results will be evaluated statistically by the Wilcoxon test and two tailed test to determine the ratio. Statistical significance will be considered at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* healthy ASA [American Society of Anaesthesiologists] class 1 patients with mandibular bilateral, symmetrical, impacted third molars indicated for extraction.

Exclusion Criteria:

* unilateral impacted and bilateral asymmetrical impacted molars;
* those who misused alcohol, had chronic pain,
* those who took narcotic drugs, beta-blockers, or any analgesic drug within 24 hours before the operation
* those with known hypersensitivity to amide types of local anesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
POSTOPERATIVE ANALGESIA EXPERIENCED BY THE PATIENTS | 5 DAYS
  THE PATIENT TO RECORD THE DURATION OF ANALGESIA AFTER SURGICAL REMOVAL OF MANDIBULAR THIRD MOLARS.

SECONDARY OUTCOMES:
NUMBER OF ORAL ANALGESICS INGESTED AFTER THE SURGICAL REMOVAL OF MANDIBULAR THIRD MOLAR TEETH. | 5 DAYS
  PATIENT WILL RECORD THE NUMBER OF ANALGESICS INGESTED IN A 5 DAY PERIOD AFTER SURGICAL REMOVAL OF MANDIBULAR THIRD MOLARS.
ADVERSE EFFECTS FROM INGESTION OF ORAL ANALGESICS | 5 DAYS
  PATIENT WILL REGISTER ANY COMPLAINTS ARISING OUT OF ORAL ANALGESIC INTAKE
DURATION OF TISSUE ANESTHESIA POSTOPERATIVELY | 1.5 TO 10 HOURS
  PATIENTS WILL RECORD THE DURATION OF TISSUE ANESTHESIA AFTER THE SURGERY